CLINICAL TRIAL: NCT04068584
Title: Evaluation of the Impact of the SMART ANGEL ™ Device on Follow-up at Home Following Major or Intermediate Outpatient Surgery: Randomized Controlled Open-label Trial
Brief Title: Evaluation of the Impact of the SMART ANGEL ™ Device on Follow-up at Home Following Major or Intermediate Outpatient Surgery
Acronym: SMART ANGEL 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Evolucare Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CIVI/2018/PC-01
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Ambulatory Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete Smart Angel (Experimental): Smat Angel application with artificial intelligence
  Interventions: Other: Smart Angel
- Basic Smart Angel (Experimental): Smat Angel application without artificial intelligence
  Interventions: Other: Smart Angel
- Control (No Intervention)

INTERVENTIONS:
Other: Smart Angel — Patient issued with a tablet with the Smart Angel application to monitor clinical signs and symptoms
  Arms: Basic Smart Angel; Complete Smart Angel

SUMMARY:
The investigators hypothesize that by monitoring and analyzing physiological parameters (heart rate, blood pressure, saturation) and well-being (pain, nausea, vomiting, comfort) the SMART ANGEL ™ device improves the quality of care after major or intermediate outpatient surgery. This active surveillance will result in a decrease in the rate of unplanned recourse (hospitalization, consultation, telephone call).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is undergoing ambulatory surgery for:

  * in orthopedics: shoulder (arthroscopy, abutment, prosthesis), hip (prosthesis, arthrolysis), knee (osteotomy, ligamentoplasty), ankle (prosthesis, ligamentoplasty) foot (hallux valgus); removal of major or multi-site equipment;
  * digestive (cholecystectomy, hernia repair, partial gastrectomy, colectomy, cleaning);
  * in gynecology (hysterectomy, oophorectomy, mastectomy, quadrantectomy, dissection, cystoplasty, sphincter);
  * in urology (total or partial resection of the prostate);
  * ENT (thyroidectomy, tonsillectomy);
  * Neurosurgery (herniated disc);
  * Vascular (stripping varix, creating fistula).
* The patient has sufficient intellectual and cognitive capacity to use the devices
* The patient must pass the test performed during the anesthesia consultation, namely:

  * open and connect the tablet,
  * activate the measurement of the blood pressure and the measurement of the oxygen saturation,
  * be connected to a 4G network

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant
* The patient is undergoing emergency or minor surgery
* Patient has a psychological class ASA 5
* Patient is non-eligible for ambulatory surgery for medical reasons (decompensated medical pathology) or social reasons according to the criteria defined by the société française anesthésie réanimation. Person lives alone or has a geographical distance from a hospital center> 30 km (or> 45 min by car).
* Patient who doesn't classify for ambulatory surgery at time of discharge

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Non-scheduled hospitalization rates between groups | Day 5
Number of non-scheduled consultations between groups | Day 5
Rates of calls with nurses between groups | Day 5
Rates of calls with doctors between groups | Day 5
Rates of unplanned prescriptions between groups | Day 5
Rates of unplanned exams between groups | Day 5

SECONDARY OUTCOMES:
Rate of complications between groups | Day 1
  % patients reported any of: nausea, vomiting, constipation, allergy, shivering, insomnia, pain, fever, sore throat, lower back pain, headache, hypotension, bradycardia, hallucination, fainting, reopening of the incision, repeated surgery, abscess, bleeding, or bruising
Rate of complications between groups | Day 2
  % patients reported any of: nausea, vomiting, constipation, allergy, shivering, insomnia, pain, fever, sore throat, lower back pain, headache, hypotension, bradycardia, hallucination, fainting, reopening of the incision, repeated surgery, abscess, bleeding, or bruising
Rate of complications between groups | Day 3
  % patients reported any of: nausea, vomiting, constipation, allergy, shivering, insomnia, pain, fever, sore throat, lower back pain, headache, hypotension, bradycardia, hallucination, fainting, reopening of the incision, repeated surgery, abscess, bleeding, or bruising
Rate of complications between groups | Day 4
  % patients reported any of: nausea, vomiting, constipation, allergy, shivering, insomnia, pain, fever, sore throat, lower back pain, headache, hypotension, bradycardia, hallucination, fainting, reopening of the incision, repeated surgery, abscess, bleeding, or bruising
Rate of complications between groups | Day 5
  % patients reported any of: nausea, vomiting, constipation, allergy, shivering, insomnia, pain, fever, sore throat, lower back pain, headache, hypotension, bradycardia, hallucination, fainting, reopening of the incision, repeated surgery, abscess, bleeding, or bruising
Rate of complications between groups | Month 1
  % patients reported any of: nausea, vomiting, constipation, allergy, shivering, insomnia, pain, fever, sore throat, lower back pain, headache, hypotension, bradycardia, hallucination, fainting, reopening of the incision, repeated surgery, abscess, bleeding, or bruising
Rate of readmission between groups | Month 1
  Yes/No
Date of return to work or other activity | 1 Month
  Dd/mm/yyyy
Patient satisfaction | Day 6
  Visual Analog Scale 0-10
Patient quality of life | 1 month
  EQ-5D-5L questionnaire taken over the phone
Difficulties in using the device | Day 5
  In-house developed usage questionnaire assessing measurement difficulties, saving errors, connection problems, problem contacting care staff
Requirement of external help in using the device | Day 5
  Description of person sought for advice
Times spent on device | Day 5
  Hours; automatically calculated by device for time used for manipulation and time for navigation
Technical errors arising | Day 5
  Automatically calculated by device

CONTACTS AND LOCATIONS:
Overall Officials: Christhophe Boisson, Study Director — CHU Nimes
Locations (24):
- France (24):
  - Polyclinique du Parc Rambot, Aix-en-Provence
  - Clinique Bonnefon, Alès
  - Centre hospitalier universitaire Amiens-Picardie, Amiens
  - Centre hospitalier D'Arles, Arles
  - Centre Hospitalier Henri Duffaut, Avignon
  - CHU Bordeaux II, Bordeaux
  - CH antoine gayraud, Carcassonne
  - Hôpital Henri-Mondor, Créteil
  - CHU Lille, Lille
  - Clinique Via Domitia, Lunel
  - Lyon Sud, Lyon
  - Hopital Nord, Marseille
  - ICM, Montpellier
  - Hopital Saint Eloi, Montpellier
  - Hôpital Lapeyronie, Montpellier
  - CHU de Nimes, Nîmes
  - Clinique des Franciscaines, Nîmes
  - Clinique Kenval, Nîmes
  - Polyclinique Grand Sud, Nîmes
  - Clinique Jouvenet, Paris
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU de Rennes, Rennes
  - CHU de Saint-Etienne, Saint-Etienne